CLINICAL TRIAL: NCT00707863
Title: fMRI and Genotype Markers of Antidepressant Side Effects and Response in Young Adults Compare to Older Adults
Brief Title: Study of Brain Response to Emotional Pictures Using a Magnetic Resonance Imaging (fMRI) While on Escitalopram
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Sponsor
Organization: Indiana University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0711-14
Record Dates: First submitted 2008-06-30; First posted 2008-07-01 (Estimated); Results first posted 2016-10-17 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-08

CONDITIONS: Major Depression
Keywords: Escitalopram; Lexapro; fMRI; pictures
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Depressed Subjects Age: 18 - 25 yrs (Other): Subjects receiving Escitalopram (trade name: Lexapro) that are in the age range of 18-25
  Interventions: Drug: Escitalopram
- Depressed Subjects Age: 16 - 50 yrs (Other): Subjects receiving Escitalopram (trade name: Lexapro) in the age range of 26-50
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — 10 mg of Escitalopram by mouth once a day for 8 weeks
  Other Names: Lexapro

SUMMARY:
The purpose of this study is to find out what parts of the brain have increased or decreased activity when people are depressed and how antidepressant medicine changes this activity in depressed patients. The genetic samples collected are to look at variation in a gene (serotonin transporter gene), which affects the functioning of the chemical serotonin in the brain

DETAILED DESCRIPTION:
This study will measure the activity in different parts of the brain, while the patients are seeing some pictures, using Magnetic Resonance Imaging (MRI) scan. For this study three MRI scans will be conducted. One before the patient begins on any medication, one during the study after 3 weeks of treatment and one after six more weeks of treatment with a standard antidepressant called Escitalopram(trade name: Lexapro).

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-50 years and able to give voluntary informed consent.
* Satisfy criteria for Major Depressive Disorder (MDD) and current depressed episode using the Mini International Neuropsychiatric Interview (M.I.N.I.).
* 17-item Hamilton Depression Rating Scale (HDRS) score > 18.
* Satisfy criteria to undergo an MRI scan based on MRI screening questionnaire.
* Able to be managed as outpatients for initial assessment and during treatment as ascertained by the following -
* Symptoms not worsening by more than 10 points on the HDRS during the course of the study.
* No danger to self or others.

Exclusion Criteria:

* Meeting DSM-IV criteria for schizophrenia, schizophreniform disorder, schizoaffective disorder, bipolar disorder, atypical psychosis, mental retardation, or organic mental (including organic mood) disorder.
* On monoamine oxidase inhibitors in the past 2 weeks.
* History of narrow angle glaucoma.
* Lack of response of the current episode of depression to two or more adequate courses of antidepressant therapy at a clinically appropriate dose for a minimum of 4 weeks or, in the judgment of the investigator, the patient meets criteria for treatment-resistant depression.
* Use of neuroleptic in the past 2 weeks.
* Use of antidepressants in the past 2 weeks. If on fluoxetine in the past, then should not have been on this medication for 4 weeks.
* Use of mood stabilizers in the past 2 weeks.
* Use of benzodiazepines in the past 2 weeks.
* Acutely suicidal or homicidal or requiring inpatient treatment.
* Meeting DSM-IV criteria for other substance dependence within the past year, except caffeine or nicotine. The criteria will be evaluated by interview and urinary toxicology screening initially and on test days.
* Use of alcohol in the past 1 week.
* No serious medical or neurological illness as assessed by physical examination and laboratory examination including CBC and blood chemistry.
* Current pregnancy or breast-feeding.
* Metallic implants.
* Previously known positive HIV blood test as reported by the subject.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2008-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Anand, M.D., Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University Adult Psychiatric Clinic, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Depressed Subjects Age: 18 - 25 Yrs | Depressed Subjects Age: 16 - 50 Yrs
Started | 6 | 11
Completed | 6 | 8
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Depressed Subjects Age: 18 - 25 Yrs | Depressed Subjects Age: 16 - 50 Yrs | Total
Number analyzed (Participants) | 6 | 11 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 11 | 17
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22 (1) | 34 (6) | 30 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 6 | 11 | 17

OUTCOME MEASURES:

1. Primary Outcome: 17-item Hamilton Depression Rating Scale (HAM-D)
Description: Standard scale for depression used in clinical trials. Range: 0 - 54. A score of 0-7 is considered to be normal. 8 - 13 mild depression. Scores of 20 or higher indicate moderate -severe depression.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Depressed Subjects Age: 18 - 25 Yrs | Depressed Subjects Age: 16 - 50 Yrs
Number analyzed (Participants) | 6 | 8
units on a scale
  Baseline 17-item HAM-D | 18 (1) | 19 (1)
  Post-8 week treatment 17-item HAM-D | 6 (3) | 6 (4)

ADVERSE EVENTS:
Groups:
- Subjects Age: 18 - 25: Subjects receiving Escitalopram (trade name: Lexapro) that are in the age range of 18-25
  Escitalopram: 10 mg of Escitalopram by mouth once a day for 8 weeks
- Subjects Age: 26 - 50: Subjects receiving Escitalopram (trade name: Lexapro) in the age range of 26-50
  Escitalopram: 10 mg of Escitalopram by mouth per day for 8 weeks
Arm/Group | Subjects Age: 18 - 25 | Subjects Age: 26 - 50
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/11
Other Adverse Events (participants affected / at risk) | 5/6 | 11/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Subjects Age: 18 - 25 (N=6) | Subjects Age: 26 - 50 (N=11)
Nervousness (Psychiatric disorders) | 1 | 3
Twitching (Musculoskeletal and connective tissue disorders) | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 3
Nausea (Gastrointestinal disorders) | 2 | 2
Diaarhea (Gastrointestinal disorders) | 1 | 1
Decreased appetite (Gastrointestinal disorders) | 4 | 5
Increased appetite (Gastrointestinal disorders) | 1 | 1
Weakness or Fatigue (Nervous system disorders) | 2 | 3
Dizziness (Nervous system disorders) | 2 | 4
Postural hypotension (Cardiac disorders) | 2 | 2
Drowsiness (Nervous system disorders) | 3 | 5
Increased sleep (Nervous system disorders) | 4 | 5
Decreased sleep (Nervous system disorders) | 2 | 6
Sweating (Skin and subcutaneous tissue disorders) | 1 | 5
Flushing (Cardiac disorders) | 0 | 1
Edema (Cardiac disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 5
Blurred vision (Eye disorders) | 0 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 7
Anorgasmia (Reproductive system and breast disorders) | 2 | 2
Increased libido (Reproductive system and breast disorders) | 0 | 0
decreased libido (Reproductive system and breast disorders) | 2 | 4
Agitation (Psychiatric disorders) | 0 | 2
Tremor (Nervous system disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 4

LIMITATIONS AND CAVEATS:
Small number of subjects were studied

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No